CLINICAL TRIAL: NCT02236169
Title: An Open-Label, Crossover, Pharmacokinetic Trial to Determine the Comparability of 84 µg Ipratropium Bromide HFA-134a Inhalation Aerosol to 84 µg ATROVENT® CFC Inhalation Aerosol, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Trial to Determine the Comparability of Ipratropium Bromide Hydrofluoroalkane (HFA)-134a Inhalation Aerosol to ATROVENT® Chlorofluorocarbon (CFC) Inhalation Aerosol, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 244.2480
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Ipratropium bromide (Experimental)
  Interventions: Drug: Ipratropium bromide HFA-134a inhalation aerosol
- ATROVENT (Active Comparator)
  Interventions: Drug: Atrovent CFC inhalation aerosol

INTERVENTIONS:
Drug: Ipratropium bromide HFA-134a inhalation aerosol
  Arms: Ipratropium bromide
Drug: Atrovent CFC inhalation aerosol
  Arms: ATROVENT

SUMMARY:
The objective of this study was to determine the pharmacokinetic comparability of 84 µg ipratropium bromide HFA-134a inhalation aerosol and 84 µg ATROVENT® CFC Inhalation Aerosol in COPD patients

ELIGIBILITY:
Inclusion Criteria:

All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

* Patients must have a stable, moderate to severe airway obstruction with an Forced Expiratory Volume in one second (FEV1) <=65% of predicted normal and FEV1 <=70% of Forced vital capacity (FVC)

  * Males: Predicted Normal FEV1 = 0.093 (height in inches)-0.032 (age)-1.343
  * Females: Predicted Normal FEV1 = 0.085 (height in inches)-0.025(age)-1.692
* Male or female age 40 years or older
* Patients must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes (20 cigarettes) per day for a year
* Patients must be able to satisfactorily administer the medication, perform pulmonary function tests (PFTs) and maintain records during the study period as required in the protocol
* All patients must sign an Informed Consent Form prior to participation in the trial (i.e., prior to pre-study washout of their usual pulmonary medications and prior to fasting for laboratory tests)

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease with may influence the results of the study or patients ability to participate in the study
* Patients with clinically relevant baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion the patient is excluded
* All patients with serum glutamic oxaloacetic transaminase (SGOT) >80 IU/L, serum glutamic pyruvic transaminase (SGPT) >80 IU/L, bilirubin >2.0 mg/dl, or creatinine >2.0 mg/dl will be excluded regardless of the clinical condition. Repeat laboratory evaluation will be not be conducted in these patients
* Patients with a history of asthma, allergic rhinitis or atopy or who have a blood eosinophil count above 600/mm3. A repeat eosinophil count will be not be conducted in these patients
* Patients with a recent (i.e., one year or less) history of myocardial infarction
* Patients with a recent history (i.e., three years or less) of cardiac failure, patients with cardiac arrhythmia requiring therapy, patients receiving any systemic beta-blockers and patients on chronic daytime oxygen therapy
* Patients with known active tuberculosis
* Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reason should be evaluated per exclusion criterion No.1
* Patients with an upper respiratory tract infection or COPD exacerbation in the 6 weeks prior to the screening visit (Visit 1) or during the baseline period
* Patients with known hypersensitivity to anticholinergic drugs
* Patients with known symptomatic prostatic hypertrophy or bladder-neck obstruction
* Patients with known narrow-angle glaucoma
* Patients who are on cromolyn sodium or nedocromil sodium
* Patients who are on antihistamines
* Pregnant or nursing women and women of childbearing potential not using a medically approved means of contraception (e.g., oral contraceptive, intrauterine devices, diaphragm or Norplant®)
* Patients who have taken an investigational drug within 1 month or 6 half-lives (whichever is longer) of the drug prior to the screening visit or patients currently enrolled in another research study
* Patients with a history of and/or active alcohol or drug abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-10; Primary Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Amount of unchanged ipratropium excreted in the urine from 0 to 24 h after a single dose | Up to 24 hours (h) after single drug administration
Amount of unchanged ipratropium excreted in the urine within 1 hour at steady state | 1h after drug administration
Amount of unchanged ipratropium excreted in the urine over the 6 h dosing interval at steady state | up to 6 h after drug administration

SECONDARY OUTCOMES:
Area under the plasma ipratropium concentration time curve at different time points | Up to 23 days after first drug administration
Peak plasma ipratropium concentration at different time points | Up to 23 days after first drug administration
Trough plasma ipratropium concentration at different time points | Up to 23 days after first drug administration
Time to peak plasma ipratropium concentrations at steady state | Up to 23 days after first drug administration
Degree of fluctuation (DF) of the plasma ipratropium concentrations | Up to 23 days after first drug administration
Area under the plasma ipratropium concentration time curve | Day 1 after first drug administration
Peak plasma ipratropium concentration | Day 1 after first drug administration
Number of patients with adverse events | Up to 23 days after first drug administration
Changes from baseline in pulse rate and blood pressure | Baseline, day 23 day after first drug administration
Number of patients with clinical significant findings in laboratory tests | Up to 23 days after first drug administration
Number of patients with clinical significant findings in physical examination | Up to 23 days after first drug administration
Number of patients with clinical significant findings in electrocardiogram (ECG) | Up to 23 days after first drug administration
Changes from test-day baseline in pulse rate and blood pressure | Up to 23 days after first drug administration